CLINICAL TRIAL: NCT01456442
Title: Short Protocol Barostat for Assessment of Anorectal Function Versus Standard Protocol Barostat in Healthy Volunteers
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: KEK-ZH-Nr. 2010-0330
Record Dates: First submitted 2011-09-26; First posted 2011-10-20 (Estimated); Last update posted 2012-11-14 (Estimated); Status verified 2012-11

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: anorectal manometry — High-resolution anorectal manometry is done under standard clinical conditions with a 10 cm catheter inserted into the rectum loaded with pressure transducers at a distance of 6 mm in the sphincter area and an attached latex balloon at the catheter tip. It will measure the length of the anal sphincter, the static pressure and the clamping pressure during at least 3 over 40 seconds sustained maneuvers according to a standardized protocol. Mean and maximum pressure increase over the resting pressure during the first 30 seconds of the squeeze and the maximum possible squeeze time will be documented. Moreover, the initial anorectal perception threshold, the perception of urge to defecate and maximum tolerable volume balloon will be documented.
  Other Names: AHRM
Device: barostat — For the barostat study a balloon will be attached to the catheter. Instead of a barostat machine a 60ml syringe and a sphygmomanometer will be connected to the catheter and the catheter will be positioned in the rectum. The balloon is then dilated gradually to assess perception, urge and discomfort threshold in relation to rectal volume.

SUMMARY:
The aim of this monocentric, prospective, non randomised study with 25 healthy volunteers is to assess anorectal function ( i.e rectal compliance and sensory thresholds) in health with a short protocol barostat versus conventional procedures (i.e. standard barostat protocol and high resolution anorectal manometry). Anorectal dysfunction is a key mechanism in the development of fecal incontinence and symptoms of obstructive defecation.

In this study volunteers will be examined - after explanation, physical examination and verification of in- and exclusion criteria - by anorectal barostat with short and standard protocol as well as by proctoscopy and endoanal ultrasound.

DETAILED DESCRIPTION:
For a coordinated anorectal function in addition to the anal sphincter the perception of rectal distension (visceral perception) and elasticity / compliance of the anorectum and stool consistency is important. A disturbed anorectal function may lead to functional defecation disorders or incontinence.

The currently available methods for measuring physiological assessment of anorectal function mostly focus on measurement of sphincter pressures, but generally provide no complete explanation for the underlying pathophysiology of defecation disorders. By voluntary contraction of the striated muscles of the external anal sphincter and puborectalis muscle defecation can be further delayed. In addition, however, other continence mechanisms play an important role.

The Group for the Study of functional gastrointestinal disorders at the Clinic for Gastroenterology at the University Hospital of Zurich has a great expertise in the establishment of new research methods such as the already in routine clinical practice used high-resolution anorectal manometry and has conducted numerous studies with anorectal Barostat. To use the results of Barostat also in everyday clinical practice in patients with defecation disorders this technique means significant simplification of the instrumental methodology and shortening of the work described in the literature. Before the simplified barostat can be used with the shortened protocol in different patient groups and clinical practice, it generally requires the validation of the technique in healthy subjects to define the range of normal values.

ELIGIBILITY:
Inclusion criteria:

* Healthy men and women between 18 and 65 years of age without gastrointestinal disease needing medical or surgical treatment.
* No medication (with the exception of occasional intake of paracetamol)
* Availability of all investigations (high resolution anorectal manometry, anorectal barostat with short and standard protocol, proctoscopy and endoanal ultrasound to assess sphincter morphology)
* Good communication with study doctor and meeting of all study requirements.
* Written consent after detailed explanation of study.

Exclusion criteria:

* Gastrointestinal symptoms especially fecal incontinence and obstructed defecation
* Structural or functional changes of upper and lower GI Tract (i.e gastric ulcer, malignancy , symptoms of IBS)
* Symptomatic or manometrically diagnosed motility disorders of the upper and lower GI tract for example anismus
* Surgery or interventions in the lower and upper GI tract (appendectomy and hernia excluded) included congenital malformations
* Pelvic radiation therapy
* Fecal incontinence, defined as involuntary loss of liquid or hard stool
* Functional defecation disorders as defined by the ROME III criteria.
* Pregnancy with history of vaginal delivery.
* Acute or chronic disease ( for example IBD)
* Malignancy
* Intake of medication one week prior to study begin. Anticoagulants and medication influencing GI motility like prokinetics, calcium channel blockers and antibiotics
* Drug or alcohol use
* Pregnancy and lactation
* Women at reproductive age will receive pregnancy testing before inclusion into study.
* Physical, mental , neurological or psychiatric conditions limiting ability to meet inclusion criteria

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2011-01; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Assessment of anorectal perception thresholds with short protocol barostat in healthy volunteers | during hospital stay, estmated 0.5 days

SECONDARY OUTCOMES:
anorectal perception thresholds in % in relation to rectal capacity assessed in ml | at time of hospital stay approx 0.5 days
  Comparison of anorectal perception thresholds and rectal capacity with the simplified barostat protocol with:
  1. the anorectal perception thresholds and rectal capacity in accordance with the standard protocol
  2. the pressure of the anal sphincter and the length at rest and during voluntary contraction,
  3. the length and the morphological integrity of the anal sphincter detected by ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: 01 Studienregister MasterAdmins, Study Director — UniversitaetsSpital Zuerich; Heiko Fruehauf, MD, Principal Investigator — University Hospital Zurich, Division of Gastroenterology and Hepatology
Locations (1):
- University Hospital Zurich, Gastroenterology and Hepatology, Zurich, Switzerland

REFERENCES:
- [Derived] Sauter M, Heinrich H, Fox M, Misselwitz B, Halama M, Schwizer W, Fried M, Fruehauf H. Toward more accurate measurements of anorectal motor and sensory function in routine clinical practice: validation of high-resolution anorectal manometry and Rapid Barostat Bag measurements of rectal function. Neurogastroenterol Motil. 2014 May;26(5):685-95. doi: 10.1111/nmo.12317. Epub 2014 Feb 12. PMID 24517865